CLINICAL TRIAL: NCT07251049
Title: Acute Infectious Encephalitis and Myelitis in Guadeloupe by New Generation Sequencing Acute Infectious Encephalitis and Myelitis in Guadeloupe by New Generation Sequencing
Brief Title: Acute Infectious Encephalitis and Myelitis in Guadeloupe by New Generation Sequencing
Acronym: EMAI-NGS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Other Study IDs: PAP_RI2_2019/10
Record Dates: First submitted 2025-11-14; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-10

CONDITIONS: Acute Encephalitis; Acute Myelitis
Keywords: Acute Infectious encephalitis; myelitis; next generation sequencing; French West Indies
MeSH Terms: conditions — Myelitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cerebrospinal fluid, blood, urinary
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Encephalitis or myelitis: Patients diagnosed with encephalitis or myelitis are defined as having an inflammatory or infectious involvement of the cerebral parenchyma or the spinal cord.

SUMMARY:
: Encephalitis or myelitis is defined as the inflammatory or infectious involvement of the cerebral parenchyma or spinal cord. When an infectious origin is suspected, the germ is not always identified. Next-generation sequencing could be used to correct an etiological diagnosis of these severe conditions in Guadeloupe. The rate of cases for which the infectious agent is not identified encourages continued diagnostic efforts, with the objective of identifying new pathogens or emerging pathogens, some of which may be more specific in the tropics.

DETAILED DESCRIPTION:
Encephalitis or myelitis is defined as the inflammatory or infectious involvement of the cerebral parenchyma or spinal cord. When an infectious origin is suspected, the germ is not always identified. In Guadeloupe, a region exposed to arboviruses, these infectious agents are among the causes of acute infectious attacks of the central nervous system. Other bacteria, parasites, or poorly known fungal agents may be responsible for these conditions. An observational study, retrospective over a period of 4 years, carried out at University Hospital of Guadeloupe, on cases of acute infectious attacks of the central nervous system, showed that the pathogen was not found in 45% of cases. Next Generation Sequencing (NGS) allows DNA or RNA sequencing faster and more accurately than other routine methods (serology / PCR). This technique could be used to correct an etiological diagnosis concerning these severe conditions in Guadeloupe, as part of a prospective study. Indeed, we find in the literature, more and more examples of patients suffering from these conditions of origin called "indeterminate", for which an etiological diagnosis is made thanks to the NGS, and sometimes a suitable curative treatment undertaken in the course of. A study of this type would be necessary to obtain exhaustive epidemiological data and to improve understanding of these severe pathologies, the consequences of which, in the short and long term, represent real public health issues. The main objective of the study is to describe, prospectively, the etiologies of acute encephalitis and myelitis at the University Hospital of Guadeloupe by carrying out diagnostic methods which may include NGS in patients without etiological diagnosis after having benefited from a first-line assessment. The secondary objectives are to describe the clinical, paraclinical and epidemiological characteristics of these conditions, and to describe long term outcomes

ELIGIBILITY:
Inclusion Criteria:

* We selected the following eligibility criteria for patients with acute encephalitis:

  * Patient of at least 28 days of life
  * With acute onset of symptoms for more than 24 hours
  * A major criterion among the following:
* a disorder of consciousness or alertness
* memory disorder
* lethargy
* modification of personal or behavioral disorder, irritability
* confusion, disorientation in time or space

  - At least two of the following minor criteria:
* temperature above 38 ° C
* new onset focal neurological deficit
* epileptic crisis
* biological abnormality of CSF (≥ 5 Leukocytes / mm3, protein ≥ 0.40 g / L)
* partial or general epileptic seizure (s) not attributable to pre-existing epileptic disease and / or a recent focal neurological symptom
* brain imaging suggestive of encephalitis, with EEG abnormalities suggestive of encephalitis

  * And absence of alternative diagnosis (intoxication, metabolic encephalopathy)
  * Persons affiliated or benefiting from a social security scheme;
  * Having given free, informed, written and signed consent by the patient or his legal representative (no later than the day of inclusion and prior to any review required by the research);
* Eligibility criteria for Acute Transverse Myelitis Patients:

  * Patient of at least 28 days of life
  * Acute onset of symptoms for more than 24 hours
  * Medullary focal abnormality, responsible for motor, sensory or autonomic symptoms
  * contrast enhancement on bone marrow MRI and / or abnormal CSF (≥ 5GB / mm3, protein uptake ≥ 0.40 g / L)
  * Evolution between nadir and maximum symptoms, less than 4 weeks
  * Persons affiliated or benefiting from a social security scheme;
  * Having given free, informed, written and signed consent by the patient or his legal representative (no later than the day of inclusion and prior to any review required by the research);

Exclusion Criteria:

* Primary vasculitis of the central nervous system or a documented specific impairment in an autoimmune condition
* Cerebral thrombophlebitis if not associated with encephalitis
* Meningitis without clinical or paraclinical argument for cerebral parenchymal involvement
* Pyogenic abscess
* Cerebral or spinal abscess
* Tumoral or hematological pathology of the central nervous system
* Toxic or metabolic encephalopathy
* Transverse myelitis with vascular or traumatic origin
* Known chronic infection with HTLV virus

Min Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with suspected acute infectious encephalitis and / or myelitis, according to the clinical and paraclinical criteria described in recommendations of the International Encephalitis Consortium in 2013 and the by the Transverse Myelitis Consortium Working Group in 2002
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-16 (Actual); Primary Completion 2028-11-16 (Estimated); Study Completion 2028-11-16 (Estimated)

PRIMARY OUTCOMES:
neurotropic pathogen | baseline, 3 month (if necessary)
  The detection of a neurotropic pathogen in the cerebrospinal fluid

SECONDARY OUTCOMES:
Neuro radiological | baseline, 3 month, 12 month
  Neuro radiological observations
Bacteriological | baseline, 15 days , 3 months
  Bacteriological observations
biochimical | baseline, 15 days, 3 months
  biochimical observations
Clinical neurological | at day 0, at hospital discharge or maximum on the 15th day (+/- 30 days), and 3 months, 12 months
  Clinical neurological examination
• Neuropsychological | 3 months, 12 months
  • Neuropsychological assessment

CONTACTS AND LOCATIONS:
Overall Officials: Hugo CHAUMONT, Doctor, Principal Investigator — CHU de la Guadeloupe
Locations (1):
- Centre Hospitalier Universitaire de la Guadeloupe, Pointe-à-Pitre, Guadeloupe, Guadeloupe

IPD SHARING:
Plan to Share IPD: No